CLINICAL TRIAL: NCT03973658
Title: Dizziness Among First Time Users of Hearing Aids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 0132-18-COM2
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-05

CONDITIONS: Dizziness; Hearing Loss
MeSH Terms: conditions — Dizziness; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First time users of hearing aids: Hearing aid fitting and usage
  Interventions: Device: Hearing aids

INTERVENTIONS:
Device: Hearing aids — Fitting of hearing aids (for the first time)

SUMMARY:
The score on the Dizziness Handicap Inventory (short version) before and after hearing aid fitting and usage will be compared

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking
* First time users of hearing aids

Exclusion Criteria:

* Using a wheelchair
* Neurological disorders
* Spine of leg surgery in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older patients using hearing aids for the first time
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (short version) score. The scale measures the degree of dizziness associated handicap as experienced by the patient. Minimun score: 0 Maximum score: 13. A higher score means better outcome. | 2 months
  The change in the score a 2 months after fitting the hearing aids

SECONDARY OUTCOMES:
Usage of hearing aids | 2 months
  The duration the participants used the hearing aids

IPD SHARING:
Plan to Share IPD: No